CLINICAL TRIAL: NCT05121701
Title: Airway Management During the Covid-19 Pandemic: A Comparison of Direct Laryngoscopy Versus Video Laryngoscopy
Brief Title: Covid-19 Pandemic and Use of Video Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Van Bölge Eğitim ve Araştırma Hastanesi (Other Government)
Responsible Party: Principal Investigator, sedef gülçin ural, Medical Doctor, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERZURUMSEHIR1
Record Dates: First submitted 2021-11-15; First posted 2021-11-16 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscopy (Active Comparator): The patients were intubated with the C-MAC PM-Karl Storz Video laryngoscope.
  Interventions: Device: Videolaryngoscope
- Laryngoscopy (Active Comparator): The patients were intubated with the Macintosh laryngoscope.
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: Videolaryngoscope — C-MAC PM-Karl Storz
  Arms: Videolaryngoscopy
Device: Macintosh Laryngoscope — Laryngoscope
  Arms: Laryngoscopy

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) causes a highly contagious infection with the highest viral load in the upper respiratory secretions. Despite using personal protective equipment, SARS-CoV-2 contamination to the healthcare personnel is possible during the airway management of infected patients. Direct laryngoscopy remains as the most common method for endotracheal intubation. Our study aimed to compare the use of video laryngoscopy with direct laryngoscopy for tracheal intubation in adult patients receiving general anesthesia for elective surgery during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Elective surgery

Exclusion Criteria:

* Intraoral or neck surgery
* gastroesophageal reflux
* delayed gastric emptying
* pregnancy
* scoliosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Intubation time | First 5 minutes of the operation
  Time from Beginning of Intubation to Full Ventilation of the Lungs

SECONDARY OUTCOMES:
Intubation Comfort | First 5 minutes of the operation
  Scale(0=bad, 1=moderate, 2=good 3=very good)
Cormack-Lehane Scoring | First 5 minutes of the operation
  Scale(1= Full view of glottis, 2=Partial view of glottis 3=Only epiglottis seen, none of glottis seen 4=Neither glottis nor epiglottis seen)

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum City Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piepho T, Fortmueller K, Heid FM, Schmidtmann I, Werner C, Noppens RR. Performance of the C-MAC video laryngoscope in patients after a limited glottic view using Macintosh laryngoscopy. Anaesthesia. 2011 Dec;66(12):1101-5. doi: 10.1111/j.1365-2044.2011.06872.x. Epub 2011 Aug 25. PMID 21883131